CLINICAL TRIAL: NCT07010887
Title: Defining the Role of Repetitive Head Impact Time Intervals in Mitigating Subconcussive Neural Injury
Brief Title: RHI Interval Effects on Brain Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); University of Rochester (Other); Boston Children's Hospital (Other); University at Buffalo (Other)
Responsible Party: Principal Investigator, Keisuke Kawata, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 24461
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-05

CONDITIONS: Repetitive Head Impacts
Keywords: Subconcussive brain injury; TBI; Soccer Heading; Time Interval

STUDY DESIGN:
Intervention Model Description: The short interval group will be assigned to undergo 16 soccer headings twice per week, with 24 hours in between each heading session. The long interval group will be assigned to undergo 16 soccer headings twice per week, with 72 hours in between each heading session.
  The control group that perform soccer kicking, instead of heading, will also have long and short intervals, identical to the heading group.
Who Masked: Outcomes Assessor
Masking Description: The blood biomarker experimentalist and lead statistician will be masked throughout the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Short Interval - heading (Experimental): Participants in the heading group will undergo 16 soccer headings, twice per week, with 24 hours in between each session.
  Interventions: Other: Short Interval
- Long Interval - heading (Experimental): Participants in the heading group will undergo 16 soccer headings, twice per week, with 72 hours in between each session.
  Interventions: Other: Long Interval
- Short Interval - kicking (Sham Comparator): Participants in the kicking-control group will undergo 16 soccer kicking, twice per week, with 24 hours in between each session.
  Interventions: Other: Short Interval
- Long Interval - kicking (Sham Comparator): Participants in the kicking-control group will undergo 16 soccer kicking, twice per week, with 72 hours in between each session.
  Interventions: Other: Long Interval

INTERVENTIONS:
Other: Short Interval — A standardized and reliable soccer heading protocol will be used for the experiment. Participants perform 16 headers or kicking with 1 header per 30 seconds. The sessions (twice per week for 4 weeks) will be separated by 24 hours.
  Arms: Short Interval - heading; Short Interval - kicking
Other: Long Interval — A standardized and reliable soccer heading protocol will be used for the experiment. Participants perform 16 headers or kicking with 1 header per 30 seconds. The sessions (twice per week for 4 weeks) will be separated by 72 hours.
  Arms: Long Interval - heading; Long Interval - kicking

SUMMARY:
Military service members frequently experience repetitive insults or impacts to the head (RHIs). The purpose of the proposed randomized controlled trial is to understand how time intervals affect neurological responses to repetitive subconcussive head impacts.

DETAILED DESCRIPTION:
This study will address whether, and to what extent, the interval of time between repetitive head impact (RHI) clusters (short, 24 hours; long, 72 hours) influences neuronal cellular, physiological, and functional integrity. We will leverage a human laboratory model of RHI to standardize and isolate the effects of RHI in the context of direction, magnitude, and frequency of head impact.

There are three aims that navigate this study:

Aim 1: To determine the effect of the interval of time between RHI clusters on neural cellular and molecular integrities through expression profiles of biofluid proteomic and transcriptomic biomarkers.

Hypotheses: Significant elevations in proteomic biomarkers will be observed acutely after experiencing RHI, and there will be cumulative increase in these biomarkers after 4 weeks of consistent exposure to RHI. The shorter interval of RHI clusters will yield greater degrees of biomarker changes as compared to the longer interval.

Aim 2: To examine the effect of the interval of time between RHI clusters on retinal and ocular-motor health, as assessed by retinal changes on optical coherence tomography (OCT), convergence, and pupillometry.

Hypotheses: A shorter interval of RHI clusters will result in altered retinal coherence and declines in convergence and choice reaction time compared to a longer interval. After 4 weeks of recurring exposure to RHI, declines in retinal and ocular-motor health will persist for 2-week post RHI exposure in the shorter-interval group, but the longer-interval group will normalize by the 2-week post-RHI follow-up.

Aim 3: To determine the influence of the interval of time between RHI clusters in neuronal network as assessed by quantitative EEG and choice reaction time.

Hypotheses: A shorter interval of RHI clusters will induce greater changes in EEG output acutely and chronically after RHI exposure, compared to the longer interval. Changes in EEG signals will persist for 2-week post RHI exposure in the shorter interval, but the changes will be normalized in the longer-interval group.

ELIGIBILITY:
Inclusion Criteria:

* Current soccer player (intercollegiate, club, intramural, recreational).
* At least 5 years of soccer heading experience (justification below).
* Ability to provide informed consent without a legally authorized representative (LAR).

Exclusion Criteria:

* Any head, neck, or face injury within the 6 months prior to enrollment, including concussions, that precludes participation in contact sports.
* Participants with eye conditions or diseases that could impact the blood vessels in the eye -such as but not limited to: glaucoma, macular degeneration, diabetic retinopathy.
* Determination that the participant is unsuitable for study entry or potentially unable to complete all aspects of the study based on the judgement of the Investigator.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Blood Biomarkers | Baseline, 24 hours following the final heading session, 14 days following the final heading session
  The primary outcome analyses will be comparing group differences (group x time interactions) in blood biomarkers, specifically NF-L (neurofilament light), phosphorylated tau (picogram per milliliter), and GFAP (glial fibrillary acidic protein; nanograms per milliliter). The aggregation of all blood biomarkers will provide a comprehensive overview of the biofluid profile of the participant following repetitive head injury.
Optical Coherence Tomography/Angiography (OCT/A) | Baseline, 24 hours following the final heading session, 14 days following the final heading session
  Retinal neural structure will be imaged in one or both eyes using high-definition spectral domain OCT, which will be acquired using a Zeiss Cirrus OCT scanner. The primary OCT variables examined will be macula CSF thickness (an indicator of the gain or loss of neurons or glia in the inner nuclear, ganglion cell and nerve fiber layer), and cup-to-disc ratio (an indicator of neurodegeneration at the optic disc). Retinal vascular structure will be acquired using the OCT angiography (OCT/A) capability of the Cirrus. The primary OCT/A variable examined will be foveal avascular zone (FAZ) area reflecting the size of the central portion of the macula which contains no blood vessels, and which increases in size with loss of capillaries in the surrounding region).
Quantitative Electroencephalography (qEEG) | Baseline, 24 hours following the final heading session, 14 days following the final heading session
  An Investigational version of the BrainScope FDA-cleared qEEG acquisition device will be used in this study. The investigational nature of the device is simply based on the code which does not produce a diagnostic result for the blinded researcher. Thus, the manufacturer's full device indications/labeling document will be the same as the FDA-cleared version. An eyes-closed resting EEG will be recorded. An FDA cleared multivariate EEG marker of concussion, the Concussion Index (CI) will be used as input for this study modeling. The CI includes measures of power (absolute and relative), mean frequency, connectivity (asymmetry, coherence, phase lag, phase synchrony), complexity (fractal dimension and scale-free activity), and information theory (entropy), across and within frequency bands. Other features of interest will be included in the EEG data set.

SECONDARY OUTCOMES:
Near Point of Convergence (NPC) | Baseline, 24 hours following the final heading session, 14 days following the final heading session
  NPC will also be assessed on the BrainScope qEEG device. The automatic NPC measurement is administered in the same manner as the manual NPC test and takes less than a minute to perform. The participant focuses on the target at arm's length and slowly brings it toward the tip of their nose. The participant is instructed to stop moving the target when they see two distinct images or when the examiner observes an outward deviation of one eye. Blurring of the image is ignored. The distance between the target and the tip of the participant's nose is recorded in centimeters (cm), digitally and accurately computed by the BrainScope automated ocular function measurement (AOFM) feature.
Pupillary Size Measurement and Reactivity | Baseline, 24 hours following the final heading session, 14 days following the final heading session
  Pupillary Size Measurement and reactivity will be measured in one or both eyes using the NeurOptics PLR-4000 pupillometer device. The eye cup of the hand-held optical scanner system is placed over the participant's eye at a right angle to their axis of vision while the user uses a touchscreen to center the participant's pupil. Once centered, the user initiates the protocol by push-button, and light pulses of 121 uW intensity and 0.80 s duration are used to stimulate pupil reflex and dilation over approximately 6 seconds. The following pupillometry metrics will be collected: initial pupil diameter (maximum), ending diameter (minimum), latency (time of onset of constriction following light stimulus), constriction velocity (average), maximum constriction velocity, dilation velocity (average) and T75 (time to reach 75% of original pupil baseline after peak constriction).
Choice Reaction Time (CRT) | Baseline, 24 hours following the final heading session, 14 days following the final heading session
  CRT will also be assessed on the BrainScope qEEG device. CRT task includes a rule-based response instruction where the participant presses the right key for one set of numbers and the left key for the other set. Participants are instructed to respond quickly and accurately.

CONTACTS AND LOCATIONS:
Overall Officials: Keisuke Kawata, PhD, Principal Investigator — Indiana University Bloomington Department of Kineseology
Locations (1):
- Indiana University School of Public Health, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marchi N, Bazarian JJ, Puvenna V, Janigro M, Ghosh C, Zhong J, Zhu T, Blackman E, Stewart D, Ellis J, Butler R, Janigro D. Consequences of repeated blood-brain barrier disruption in football players. PLoS One. 2013;8(3):e56805. doi: 10.1371/journal.pone.0056805. Epub 2013 Mar 6. PMID 23483891
- [Background] Kawata K, Rubin LH, Takahagi M, Lee JH, Sim T, Szwanki V, Bellamy A, Tierney R, Langford D. Subconcussive Impact-Dependent Increase in Plasma S100beta Levels in Collegiate Football Players. J Neurotrauma. 2017 Jul 15;34(14):2254-2260. doi: 10.1089/neu.2016.4786. Epub 2017 Apr 27. PMID 28181857
- [Background] Puvenna V, Brennan C, Shaw G, Yang C, Marchi N, Bazarian JJ, Merchant-Borna K, Janigro D. Significance of ubiquitin carboxy-terminal hydrolase L1 elevations in athletes after sub-concussive head hits. PLoS One. 2014 May 7;9(5):e96296. doi: 10.1371/journal.pone.0096296. eCollection 2014. PMID 24806476
- [Background] Oliver JM, Jones MT, Kirk KM, Gable DA, Repshas JT, Johnson TA, Andreasson U, Norgren N, Blennow K, Zetterberg H. Serum Neurofilament Light in American Football Athletes over the Course of a Season. J Neurotrauma. 2016 Oct 1;33(19):1784-1789. doi: 10.1089/neu.2015.4295. Epub 2016 Mar 16. PMID 26700106
- [Background] Oliver JM, Anzalone AJ, Stone JD, Turner SM, Blueitt D, Garrison JC, Askow AT, Luedke JA, Jagim AR. Fluctuations in blood biomarkers of head trauma in NCAA football athletes over the course of a season. J Neurosurg. 2018 May 29;130(5):1655-1662. doi: 10.3171/2017.12.JNS172035. Print 2019 May 1. PMID 29807487
- [Background] Shahim P, Zetterberg H, Tegner Y, Blennow K. Serum neurofilament light as a biomarker for mild traumatic brain injury in contact sports. Neurology. 2017 May 9;88(19):1788-1794. doi: 10.1212/WNL.0000000000003912. Epub 2017 Apr 12. PMID 28404801
- [Background] Joseph JR, Swallow JS, Willsey K, Lapointe AP, Khalatbari S, Korley FK, Oppenlander ME, Park P, Szerlip NJ, Broglio SP. Elevated markers of brain injury as a result of clinically asymptomatic high-acceleration head impacts in high-school football athletes. J Neurosurg. 2018 Jul 3;130(5):1642-1648. doi: 10.3171/2017.12.JNS172386. Print 2019 May 1. PMID 29966462
- [Background] Tierney GJ, Higgins B. The incidence and mechanism of heading in European professional football players over three seasons. Scand J Med Sci Sports. 2021 Apr;31(4):875-883. doi: 10.1111/sms.13900. Epub 2021 Jan 18. PMID 33280186
- [Background] Peek K, Vella T, Meyer T, Beaudouin F, McKay M. The incidence and characteristics of purposeful heading in male and female youth football (soccer) within Australia. J Sci Med Sport. 2021 Jun;24(6):603-608. doi: 10.1016/j.jsams.2020.12.010. Epub 2020 Dec 26. PMID 33414022
- [Background] Russell ER, Mackay DF, Stewart K, MacLean JA, Pell JP, Stewart W. Association of Field Position and Career Length With Risk of Neurodegenerative Disease in Male Former Professional Soccer Players. JAMA Neurol. 2021 Sep 1;78(9):1057-1063. doi: 10.1001/jamaneurol.2021.2403. PMID 34338724
- [Background] Mackay DF, Russell ER, Stewart K, MacLean JA, Pell JP, Stewart W. Neurodegenerative Disease Mortality among Former Professional Soccer Players. N Engl J Med. 2019 Nov 7;381(19):1801-1808. doi: 10.1056/NEJMoa1908483. Epub 2019 Oct 21. PMID 31633894
- [Background] Kawata K, Tierney R, Phillips J, Jeka JJ. Effect of Repetitive Sub-concussive Head Impacts on Ocular Near Point of Convergence. Int J Sports Med. 2016 May;37(5):405-10. doi: 10.1055/s-0035-1569290. Epub 2016 Feb 9. PMID 26859643